CLINICAL TRIAL: NCT06500208
Title: An Open-label, One-arm Phase II Study of Adebrelimab Combined With Neoadjuvant Chemotherapy for High-risk, Early-stage and Locally Advanced Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative (ER+/HER2-) Breast Cancer.
Brief Title: Neoadjuvant Adebrelimab and Chemotherapy in High-rish ER+/HER2- BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC-2402
Record Dates: First submitted 2024-07-06; First posted 2024-07-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; ER+/HER2-; neoadjuvant; Adebrelimab
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab and chemotherapy (Experimental): Adebrelimab 1200 mg Q3W combined with nab-paclitaxel (100 mg/m2 Q1W) for 4 cycles followed by epirubicin (90 mg/m2) and cyclophosphamide (600 mg/m2) Q3W for 4 cycles.
  Interventions: Drug: Adebrelimab combined with nab-paclitaxel, epirubicin and cyclophosphamide

INTERVENTIONS:
Drug: Adebrelimab combined with nab-paclitaxel, epirubicin and cyclophosphamide — Adebrelimab 1200mg i.v. q3w combined with nab-paclitaxel 100mg/m2 qw*12w followed by epirubicin 90mg/m2 and cyclophosphamide 600mg/m2 q3w for 4 cycles

SUMMARY:
Investigators plan to conduct a single-arm clinical study of adebelimab, a novel PD-L1 inhibitor, in the neoadjuvant treatment of early or locally advanced high-risk ER+/HER2- breast cancer, to explore whether the addition of immune checkpoint inhibitors to traditional neoadjuvant chemotherapy can improve the pathologic complete response rate (pCR) of patients, evaluate its therapeutic safety, and further analyze the biomarkers of the efficacy of neoadjuvant immunotherapy for ER+/HER2- breast cancer, so as to support the clinical application of the drug.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as unilateral primary invasive breast cancer with a) cT1c-T2N1-3 or cT3-4N0-3, b) Tumor Grade 3 or Grade 2 with PR- or Ki67 > 20%;
* IHC ER expression ≥1%; IHC HER2 0 or 1+; IHC HER2 2+ and no amplification in FISH test;
* At least one measurable lesion according to RECIST 1.1;
* Available core needle biopsy samples for PD-L1 status testing;
* ECOG 0 or 1 within 10 days prior to initiation of treatment;
* Not currently pregnant or breastfeeding, agree to strict contraception during treatment and at least 6 months after last dose;
* Intact hematologic, liver, renal and heart functions;
* Signed written informed consent.

Exclusion Criteria:

* Bilateral invasive breast cancer or Stage IV breast cancer;
* Severe heart disease;
* Diagnosed as immune deficiency or receiving systemic steroid therapy or any form of immuno-suppressive therapy within 7 days prior to the first dose of treatment;
* Had active autoimmune diseases requiring systemic therapy within the past 2 years;
* Severe systemic infections or other serious medical conditions;
* Other malignant tumors in the past 5 years, except for cured carcinoma in situ of the cervix and skin cancer without melanoma;
* History of HIV infection;
* Active HBV or HCV infection;
* Known allergies or intolerance to the therapeutic drug or its excipients;
* History of application of any immunotherapy targeting PD-1/PD-L1/T cell receptors;
* Judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate | up to 8 months, after patients complete surgery
  pathological complete response rate: No invasive residual disease in surgical specimen of breast and axillary lymph nodes

SECONDARY OUTCOMES:
ORR | up to 8 months, after patients complete surgery
  Objective Response Rate: patients achieving partial response and complete response during treatment
Incidence of adverse events (Safety) | up to 8 months, after patients complete surgery
  adverse events of patients receiving at least one cycle of treatment
pCR rate in PD-L1 CPS≥1 subgroup | up to 8 months, after patients complete surgery
  pathological complete response rate in patients with PD-L1 CPS score ≥1

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No